CLINICAL TRIAL: NCT05247801
Title: Safe Use of Medication at Home by Caregivers. Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Servicio Aragonés de Salud (SALUD) (Unknown); Fondo de Investigación en Salud (FIS) (Unknown); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunidad Valenciana (Unknown); Hospital General de Elda (Other); Servicio Navarro de Salud - Osasunbidea (Unknown); Hospital Universitari Sant Joan d'Alacant (Unknown); Hospital Universitario San Cecilio (Unknown); Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PI21/00646
Record Dates: First submitted 2022-01-21; First posted 2022-02-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Caregivers of Multi-pathological and Polypharmacy Adults
Keywords: Medication Errors; Patient Safety; Psychoeducational Intervention; Risk Management; Health Literacy

STUDY DESIGN:
Intervention Model Description: Participants. Caregivers of multi-pathological and polypharmacy patients (Barthel equal to or lower than 55). Recruitment will be carried out by simple randomization based on the diaries of patients seen in the last 18 months in the collaborating centers.
  Intervention. Psychoeducational intervention based on virtual reality aimed at increasing self-efficacy and health literacy in medication use.
  Procedure. By simple randomization, participants will be assigned to one of the two groups (control or experimental) after giving their informed consent. They will not know to which group they belong.
  Treatments. The subjects in the control group will use a dosing device and will receive information on how to use it to avoid medication errors. The experimental group will receive the psychoeducational intervention and the same medication device. The experimental group will receive the psychoeducational intervention. Intervention period: 15 days. Follow-up: 6 months.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Psychoeducational Intervention) (Experimental): Seventy one caregivers of multi-pathological and polypharmacy patients will receive psychoeducational intervention based on virtual reality and a dosing device for safer medication use at home. The intervention will be developed in a previous project phase using a mixed methodology (observational study and qualitative techniques). The intervention will be group-based and consist of motivational discussions and a review of audiovisual materials to promote self-efficacy and health literacy on the safe use of medication at home (most frequent errors, preventive strategies, etc.). Study period: 15 days intervention and follow-up 6 months.
  Interventions: Behavioral: Psychoeducational intervention for safe medication use at home + Medication dosing device
- Control Group (Dosing Device) (Active Comparator): The 71 subjects assigned to the control group will use a medication dosing device and will receive information on how to use it for medication errors. Study period: 15 days intervention and follow-up 6 months.
  Interventions: Device: Medication dosing device

INTERVENTIONS:
Behavioral: Psychoeducational intervention for safe medication use at home + Medication dosing device — The intervention is yet to be defined. Psychoeducational intervention based on virtual reality, demonstrations, and psychoeducational content using virtual reality. Contents:
  Most frequent medication errors at home. Approaches to risk management in the home. Correct use of the most common medications in different patient profiles. Strategies to avoid medication errors. Guidance to alleviate the burden of responsibility suffered by women as a result of the gender bias derived from assuming the caregiver role.
  Other.
  Arms: Experimental Group (Psychoeducational Intervention)
Device: Medication dosing device — Use of medication dosing device.
  Arms: Control Group (Dosing Device)

SUMMARY:
Experimental study to test the effectiveness of a psychoeducational intervention using virtual reality, aimed at caregivers of multi-pathological and polypharmacy persons to promote safer medication use at home. Experimental design with two groups (experimental and control), pre-post measures, and participants assignment to groups by simple randomization.

Null hypothesis. There will be no differences in the frequency of medication errors at home, the severity of the consequences of medication errors, perceived self-efficacy, and health literacy between caregivers using a dosing device (control group) and caregivers using a dosing device with the reinforcement of a psychoeducational intervention designed ad hoc (experimental group).

DETAILED DESCRIPTION:
Background. Population aging is leading to an increase in the number of multi-pathological and polymedicated patients. These patients are at increased risk of suffering adverse events due to medication errors (ME), especially if Barthel≤55. The management of their medication places an added burden of stress on those who assume responsibility for their care. This task, due to the existing gender gap, falls more often on women.

Objective. To promote the safe use of medication in the home by those who assume the role of caregivers of these patients.

Method. Mixed research study. First: Nominal groups (N=128) and survey (N=1255) to design a psychoeducational intervention aimed at caregivers based on the identification of ME, its causes and consequences, and risk factors that contribute to ME. Second: Single-subject experimental design (two groups, experimental and control, with pre-post measures) to determine the effectiveness of the psycho-educational intervention (n=142).

Setting. Primary care centers and caregivers' associations and training schools in Alicante, Granada, Madrid, Pamplona, Seville, and Zaragoza.

Expected results. Identify critical elements for medication risk management in the home by caregivers. Low-cost psycho-educational intervention for safer use of medication adjusted to the possible different needs of male and female caregivers. The transfer of results will be mainly oriented to reinforce the action carried out by nursing and caregivers' training schools.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of multi-pathological and polypharmacy patients (Barthel equal to or less than 55).
* Residence in Alicante, Granada, Madrid, Pamplona, Seville, or Zaragoza (in the patient's home or the family member's home).
* At patient's charge for at least six months during the year.

Exclusion Criteria:

* Caregivers of patients who are institutionalized a minimum of 3 months per year.
* Caregivers with experience of more than six months in the use of medication dosing devices.
* Health education/profession.
* Filing of a property claim in the last 5 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 142 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Frequency of Medication Errors after the intervention (6 months later). | Pre-intervention measure (6 months prior). Post-intervention measure (last 6 months).
  The number of medication errors, type, and consequences (adverse events and consumption of healthcare resources to mitigate the effect of the error). Self-reported measure. Pre-intervention measure (6 months prior). Post-intervention measure (last 6 months).
Change from Baseline Health Literacy after the intervention (6 months later). | Pre- and post-intervention measurement (6 months time lapse).
  Health Literacy validated questionnaire.
Change from Baseline Therapeutic Adherence after the intervention (12 months later). | Pre- and post-intervention measurement (12 months time lapse).
  Therapeutic Adherence validated questionnaire.
Change from Baseline Locus of Control after the intervention (12 months later). | Pre- and post-intervention measurement (12 months time lapse).
  Locus of Control Test - Abridged.
Change from Baseline Self-efficacy after the intervention (12 months later). | Pre- and post-intervention measurement (12 months time lapse).
  Adaptation of the Family Caregiver Activation in Transitions (FCAT) Tool (Coleman et al., 2015).
Perceived usefulness of the information provided at the time of intervention completion. | Post-intervention measure (15 days after the start of the intervention).
  Ad hoc survey
Perceived usefulness of the information provided after 3 months from the end of the intervention. | Post-intervention measure (after 3 months).
  Ad hoc survey
Perceived usefulness of the information provided after 6 months from the end of the intervention. | Post-intervention measure (after 6 months).
  Ad hoc survey
Perceived usefulness of the information provided after 12 months from the end of the intervention. | Post-intervention measure (after12 months).
  Ad hoc survey
Family Caregivers' Experience at the time of intervention completion. | Post-intervention measure (15 days after the start of the intervention).
  The Measure of the Family Caregivers' Experience (Guilabert et al., 2018).
Family Caregivers' Experience after 3 months from the end of the intervention. | Post-intervention measure (after 3 months).
  The Measure of the Family Caregivers' Experience (Guilabert et al., 2018).
Family Caregivers' Experience after 6 months from the end of the intervention. | Post-intervention measure (after 6 months).
  The Measure of the Family Caregivers' Experience (Guilabert et al., 2018).
Family Caregivers' Experience after 12 months from the end of the intervention. | Post-intervention measure (after 6 months).
  The Measure of the Family Caregivers' Experience (Guilabert et al., 2018).

CONTACTS AND LOCATIONS:
Overall Officials: José Joaquín Mira, Ph.D., Principal Investigator — Univ. Miguel Hernández; Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la CV
Locations (1):
- Miguel Hernández University, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
The databases, without identification and code registration, will be available at OSF (Center for Open Science) for access by the scientific community. the scientific community.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Six months after the data collecting.
Access Criteria: Data repository is available for the scientific community.

REFERENCES:
- [Background] Tinetti ME, Fried TR, Boyd CM. Designing health care for the most common chronic condition--multimorbidity. JAMA. 2012 Jun 20;307(23):2493-4. doi: 10.1001/jama.2012.5265. No abstract available. PMID 22797447
- [Background] Haro JM, Tyrovolas S, Garin N, Diaz-Torne C, Carmona L, Sanchez-Riera L, Perez-Ruiz F, Murray CJ. The burden of disease in Spain: results from the global burden of disease study 2010. BMC Med. 2014 Dec 5;12:236. doi: 10.1186/s12916-014-0236-9. PMID 25480438
- [Background] Masana L. [Long-term informal care in Spain: challenges, views and solutions]. Salud Colect. 2017 Apr-Jun;13(2):337-352. doi: 10.18294/sc.2017.1237. Spanish. PMID 28832828
- [Background] Heckel L, Fennell KM, Mohebbi M, Byrnes M, Livingston PM. Demographic characteristics, call details and psychosocial support needs of the family/friends of someone diagnosed with cancer who access Australian Cancer Council telephone information and support services. Eur J Oncol Nurs. 2017 Jun;28:86-91. doi: 10.1016/j.ejon.2017.03.007. Epub 2017 Apr 6. PMID 28478861
- [Background] Park M, Choi S, Lee SJ, Kim SH, Kim J, Go Y, Lee DY. The roles of unmet needs and formal support in the caregiving satisfaction and caregiving burden of family caregivers for persons with dementia. Int Psychogeriatr. 2018 Apr;30(4):557-567. doi: 10.1017/S104161021700196X. Epub 2017 Sep 28. PMID 28956524
- [Background] Guilabert M, Amil P, Gonzalez-Mestre A, Gil-Sanchez E, Vila A, Contel JC, Ansotegui JC, Solas O, Bacigalupe MT, Fernandez-Cano P, Arteagoitia M, Mira JJ. The Measure of the Family Caregivers' Experience. Int J Environ Res Public Health. 2018 Sep 18;15(9):2040. doi: 10.3390/ijerph15092040. PMID 30231535
- [Background] Look KA, Stone JA. Medication management activities performed by informal caregivers of older adults. Res Social Adm Pharm. 2018 May;14(5):418-426. doi: 10.1016/j.sapharm.2017.05.005. Epub 2017 May 16. PMID 28528023
- [Background] Panagioti M, Khan K, Keers RN, Abuzour A, Phipps D, Kontopantelis E, Bower P, Campbell S, Haneef R, Avery AJ, Ashcroft DM. Prevalence, severity, and nature of preventable patient harm across medical care settings: systematic review and meta-analysis. BMJ. 2019 Jul 17;366:l4185. doi: 10.1136/bmj.l4185. PMID 31315828
- [Background] Mira JJ, Lorenzo S, Guilabert M, Navarro I, Perez-Jover V. A systematic review of patient medication error on self-administering medication at home. Expert Opin Drug Saf. 2015 Jun;14(6):815-38. doi: 10.1517/14740338.2015.1026326. Epub 2015 Mar 16. PMID 25774444
- [Background] Mira JJ, Navarro IM, Guilabert M, Aranaz J. [Frequency of medication errors by patients]. Rev Panam Salud Publica. 2012 Feb;31(2):95-101. doi: 10.1590/s1020-49892012000200001. Spanish. PMID 22522870
- [Background] Mira JJ, Martinez-Jimeno L, Orozco-Beltran D, Iglesias-Alonso F, Lorenzo S, Nuno R, Perez P, Toro N, Perez-Jover V, Gil-Guillen V. What older complex chronic patients need to know about their everyday medication for safe drug use. Expert Opin Drug Saf. 2014 Jun;13(6):713-21. doi: 10.1517/14740338.2014.916272. Epub 2014 May 12. PMID 24821193
- [Background] SCHWARTZ D, WANG M, ZEITZ L, GOSS ME. Medication errors made by elderly, chronically ill patients. Am J Public Health Nations Health. 1962 Dec;52(12):2018-29. doi: 10.2105/ajph.52.12.2018. No abstract available. PMID 13987359
- [Background] Grossman MR, Zak DK, Zelinski EM. Mobile Apps for Caregivers of Older Adults: Quantitative Content Analysis. JMIR Mhealth Uhealth. 2018 Jul 30;6(7):e162. doi: 10.2196/mhealth.9345. PMID 30061093
- [Background] Sala-Gonzalez M, Perez-Jover V, Guilabert M, Mira JJ. Mobile Apps for Helping Informal Caregivers: A Systematic Review. Int J Environ Res Public Health. 2021 Feb 10;18(4):1702. doi: 10.3390/ijerph18041702. PMID 33578819
- [Background] Schwappach DL. Review: engaging patients as vigilant partners in safety: a systematic review. Med Care Res Rev. 2010 Apr;67(2):119-48. doi: 10.1177/1077558709342254. Epub 2009 Aug 11. PMID 19671916
- [Background] Smith F, Francis SA, Gray N, Denham M, Graffy J. A multi-centre survey among informal carers who manage medication for older care recipients: problems experienced and development of services. Health Soc Care Community. 2003 Mar;11(2):138-45. doi: 10.1046/j.1365-2524.2003.00415.x. PMID 14629216
- [Background] Alsaeed D, Jamieson E, Gul MO, Smith FJ. Challenges to optimal medicines use in people living with dementia and their caregivers: A literature review. Int J Pharm. 2016 Oct 30;512(2):396-404. doi: 10.1016/j.ijpharm.2015.12.050. Epub 2015 Dec 22. PMID 26721728
- [Background] Hodgkinson B, Koch S, Nay R, Nichols K. Strategies to reduce medication errors with reference to older adults. Int J Evid Based Healthc. 2006 Mar;4(1):2-41. doi: 10.1111/j.1479-6988.2006.00029.x. PMID 21631752
- [Background] Appel L, Appel E, Bogler O, Wiseman M, Cohen L, Ein N, Abrams HB, Campos JL. Older Adults With Cognitive and/or Physical Impairments Can Benefit From Immersive Virtual Reality Experiences: A Feasibility Study. Front Med (Lausanne). 2020 Jan 15;6:329. doi: 10.3389/fmed.2019.00329. eCollection 2019. PMID 32010701
- [Background] Oh-Park M, Doan T, Dohle C, Vermiglio-Kohn V, Abdou A. Technology Utilization in Fall Prevention. Am J Phys Med Rehabil. 2021 Jan 1;100(1):92-99. doi: 10.1097/PHM.0000000000001554. PMID 32740053
- [Background] Brydon M, Kimber J, Sponagle M, MacLaine J, Avery J, Pyke L, Gilbert R. Virtual Reality as a Tool for Eliciting Empathetic Behaviour in Carers: An Integrative Review. J Med Imaging Radiat Sci. 2021 Sep;52(3):466-477. doi: 10.1016/j.jmir.2021.04.005. Epub 2021 May 20. PMID 34023219